CLINICAL TRIAL: NCT05940298
Title: SPECT Imaging of Gastrin Releasing Peptide Receptors Using Labeled Technetium-99m DB8 ([99mTc]Tc- DB8) in Prostate Cancer and Breast Cancer Patients
Brief Title: Molecular Imaging of Gastrin Releasing Peptide Receptors Using Labeled Technetium-99m DB8
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: [99mTc]Tc- DB8
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancer; Breast Cancer
Keywords: Prostate cancer; Breast cancer; Gastrin releasing peptide receptors; [99mTc]Tc-DB8; SPECT
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prostate cancer (Experimental): At least five (5) evaluable subjects with prostate cancer
  Interventions: Drug: Intravenous injection of [99mTc]Tc-DB8
- Breast cancer (Experimental): At least five (5) evaluable subjects with breast cancer
  Interventions: Drug: Intravenous injection of [99mTc]Tc-DB8

INTERVENTIONS:
Drug: Intravenous injection of [99mTc]Tc-DB8 — One single intravenous injection of [99mTc]Tc-DB8, followed by gamma camera imaging after 2, 4, 6 and 24 hours.
  Other Names: [99mTc]Tc-DB8

SUMMARY:
The study should evaluate the biological distribution of 99mTc-DB8 in patients with prostate cancer and breast cancer.

The primary objective are:

1. To assess the distribution of [99mTc]Tc- DB8 in normal tissues and tumors at different time intervals.
2. To evaluate dosimetry of [99mTc]Tc- DB8.
3. To study the safety and tolerability of the drug [99mTc]Tc- DB8 after a single injection in a diagnostic dosage.

The secondary objective are:

1. To compare the obtained [99mTc]Tc- DB8 SPECT imaging results with the data of CT and/or MRI and/or ultrasound examination and immunohistochemical (IHC) studies in prostate cancer and breast cancer patients.

DETAILED DESCRIPTION:
The overall goal is to study the effectiveness of SPECT imaging prostate cancer and breast cancer patients Using technetium-99m labeled DB8.

Phase I of the study:

Biodistribution of 99mTc-DB8 in patients with prostate cancer and breast cancer.

The main objectives of the study:

1. To evaluate the distribution of 99mTc-DB8 in normal tissues and tumors in patients with prostate cancer and breast cancer at different time intervals.
2. To evaluate dosimetry of 99mTc-DB8 based on the pharmacokinetic parameters of the drug after a single intravenous administration.
3. To study the safety of use and tolerability of the drug 99mTc-DB8 after a single intravenous administration in a diagnostic dosage.

Additional research tasks:

1. To conduct a comparative analysis of the diagnostic information obtained in the visualization of prostate cancer and breast cancer by SPECT using 99mTc-DB8 with data obtained by CT and/or MRI and/or ultrasound examination and immunohistochemical (IHC) research of postoperative material.

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labeled tracer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Clinical and radiological diagnosis of prostate cancer and breast cancer with histological verification.
* White blood cell count: > 2.0 x 10^9/L
* Haemoglobin: > 80 g/L
* Platelets: > 50.0 x 10^9/L
* Bilirubin =< 2.0 times Upper Limit of Normal
* Serum creatinine: Within Normal Limits
* Blood glucose level not more than 5.9 mmol/L
* A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Active current autoimmune disease or history of autoimmune disease
* Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
* Known HIV positive or chronically active hepatitis B or C
* Administration of other investigational medicinal product within 30 days of screening
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-03 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body [99mTc]Tc-DB8 uptake value (%) | 24 hours
  Whole-body [99mTc]Tc-DB8 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT-based [99mTc]Tc-DB8 value in tumor lesions (counts) | 6 hours
  [99mTc]Tc-DB8 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts
SPECT-based [99mTc]Tc-DB8 background uptake value (counts) | 6 hours
  Focal uptake of [99mTc]Tc-DB8 in the regions without pathological findings will be assessed with SPECT and measured in counts
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of [99mTc]Tc-DB8 uptake coinciding with tumor lesions (counts) will be divided by the value of [99mTc]Tc-DB8 uptake coinciding with the regions without pathological findings (counts)

SECONDARY OUTCOMES:
Safety attributable to [99mTc]Tc-DB8 injections (physical findings) | 24 hours
  The safety attributable to [99mTc]Tc-DB8 injections will be evaluated based on the assessments of physical examination, vital signs, and ECG (percent of cases with abnormal findings relative to baseline).
Safety attributable to [99mTc]Tc-DB8 injections (laboratory tests) | 24 hors
  The safety attributable to [99mTc]Tc-DB8 injections will be evaluated based on the blood and urine laboratory tests (percent of cases with abnormal findings relative to baseline).
Safety attributable to [99mTc]Tc-DB8 injections (incidence of adverse events) | 24 hours
  The safety attributable to [99mTc]Tc-DB8 injections will be evaluated based on the rate of adverse events (percent).
Safety attributable to [99mTc]Tc-DB8 injections (concomitant medication) | 24 hours
  The safety attributable to [99mTc]Tc-DB8 injections will be evaluated based on the rate of administration of concomitant medication (percent).

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD,Prof, Principal Investigator — TomskNRMC Tomsk, Russia
Locations (1):
- TomskNRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: No